CLINICAL TRIAL: NCT00956410
Title: An Open-label Extension to a 52-week, Multi-center, Randomized, Double-blind, Placebo-controlled, Parallel Group Study in Patients With Alzheimer's Disease to Investigate the Safety and Tolerability of Repeated Subcutaneous Injections of CAD106
Brief Title: To Investigate the Safety and Tolerability of Repeated Subcutaneous Injections of CAD106 in Alzheimer's Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCAD106A2201E1
Record Dates: First submitted 2009-08-10; First posted 2009-08-11 (Estimated); Last update posted 2020-02-11 (Actual); Status verified 2011-11

CONDITIONS: Alzheimer Disease
Keywords: Active immunization; Alzheimer disease; Antibody; Central Nervous System Diseases; Neurodegenerative diseases; Vaccine
MeSH Terms: conditions — Alzheimer Disease; Central Nervous System Diseases; Neurodegenerative Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CAD106 (Experimental)
  Interventions: Biological: CAD106

INTERVENTIONS:
Biological: CAD106

SUMMARY:
This study will evaluate the safety and tolerability of repeated subcutaneous injections of CAD106 in patients with Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have completed the Core study with no significant safety concerns

Exclusion Criteria:

* Diagnosis of other neurodegenerative disease and/or psychiatric disorders (with the exception of successfully treated depression).
* Diagnosis or presence of an active, uncontrolled seizure disorder and/or cerebrovascular disease.
* diagnosis or presence of an active autoimmune and/or with an acute or chronic inflammation.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2009-09; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Safety/tolerability assessments at multiple timepoints including but not limited to screening, and through to the end of the study to week 66. | 66 weeks

SECONDARY OUTCOMES:
Immune response, cognitive and functional assessments at multiple timepoints including but not limited to baseline and through to the end of the study to week 66. | 66 weeks
Evaluate the antibody response after 4 additional injections in the Extension study in patients initially treated with CAD106 in the Core study. | 66 weeks
Collect long-term safety information through SAEs collection for two years after completion of the core study, CAD106A2201, or extension study, CAD106A2201E1. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (4):
- Novartis Investigative Site, Bordeaux, France
- Novartis Investigative Site, Stockholm, Sweden
- Novartis Investigative Site, Basel, Switzerland
- Novartis Investigative Site, Southampton, United Kingdom

REFERENCES:
- [Derived] Farlow MR, Andreasen N, Riviere ME, Vostiar I, Vitaliti A, Sovago J, Caputo A, Winblad B, Graf A. Long-term treatment with active Abeta immunotherapy with CAD106 in mild Alzheimer's disease. Alzheimers Res Ther. 2015 Apr 27;7(1):23. doi: 10.1186/s13195-015-0108-3. eCollection 2015. PMID 25918556